CLINICAL TRIAL: NCT00719550
Title: A Multicenter, Double-Blind, 3-Arm, Phase 1b/2 Study in Subjects With Unresectable Locally Advanced or Metastatic Gastric or Esophagogastric Junction Adenocarcinoma to Evaluate the Safety and Efficacy of First-line Treatment With Epirubicin, Cisplatin, and Capecitabine(ECX) Plus AMG 102
Brief Title: AMG 102 Plus ECX for Unresectable Locally Advanced or Metastatic Gastric or Esophagogastric Junction Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20060317
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Esophagogastric Junction Adenocarcinoma; Gastric Cancer; Esophageal Cancer
Keywords: Locally Advanced; Metastatic
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Epirubicin; rilotumumab; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Phase 2 Arm C (Placebo Comparator): AMG 102 placebo plus ECX
  Interventions: Drug: Capecitabine; Drug: Epirubicin; Drug: Cisplatin; Drug: Placebo
- Phase 1b (Other): Phase 1b dose study with open-labe AMG 102 at 15mg/kg de-escalating to 7.5mg/kg and 5mg/kg if needed.
  Interventions: Drug: Capecitabine; Drug: Epirubicin; Drug: AMG 102; Drug: Cisplatin
- Phase 2 Arm B (Active Comparator): AMG 102 at 7.5mg/kg plus ECX
  Interventions: Drug: Capecitabine; Drug: Epirubicin; Drug: AMG 102; Drug: Cisplatin
- Phase 2 Arm A (Active Comparator): AMG 102 at 15mg/kg plus ECX
  Interventions: Drug: Capecitabine; Drug: Epirubicin; Drug: AMG 102; Drug: Cisplatin

INTERVENTIONS:
Drug: Capecitabine — Administered at 625mg/m2 BID orally every day while on study.
  Other Names: Xeloda
Drug: Epirubicin — Administered day 1 of each cycle at 50mg/m2 IV.
Drug: AMG 102 — Investigation product to be given at 15mg/kg, 7.5mg/kg, or 5mg/kg depending on assignment.
  Arms: Phase 1b; Phase 2 Arm A; Phase 2 Arm B
Drug: Cisplatin — Administered day 1 of each cycle at 60mg/m2 IV.
Drug: Placebo — AMG 102 placebo will be provided in similar vials as clear, colorless, sterile protein-free solution
  Arms: Phase 2 Arm C

SUMMARY:
Study Phase: 1b/2 Indication: Previously untreated subjects with unresectable locally advanced or metastatic gastric or esophagogastric junction adenocarcinoma.

Primary Objective(s):

Part 1: To identify safe dose levels of AMG 102, up to 15 mg/kg Q3W, to combine with ECX.

Part 2 (phase 2-double-blind): To estimate with pre-specified precision the effect of the addition of AMG 102 to ECX on progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed unresectable locally advanced or metastatic gastric or esophagogastric junction (EGJ) adenocarcinoma; tumors of the distal esophagus within 5 cm of the EGJ are eligible
* ECOG performance status 0 or 1
* Male or female ≥ 18 years of age

Exclusion Criteria:

* Previous systemic therapy (chemotherapy or biologic therapy) for locally advanced or metastatic gastric or esophagogastric adenocarcinoma
* Less than 6 months have elapsed from completion of prior neoadjuvant or adjuvant chemotherapy or chemoradiotherapy.
* Subjects with resectable disease or suitable for definitive chemoradiation
* Subjects with persistent gastric outlet obstruction, complete dysphagia or feeding jejunostomy
* Tumors of squamous cell histology
* Known central nervous system metastases
* Clinically significant upper gastro-intestinal bleeding ≤ 30 days prior to enrollment or randomization
* Serious or non-healing wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS), as measured by RECIST per local review | Subjects coming off study will be contacted by telephone or at routine clinic visits approximately every 3 months until 36 months from date the last subject is randomized into the study.

SECONDARY OUTCOMES:
Overall survival, objective response rate, disease control rate, time to response (for responders only), and duration of response (for responders only). | Subjects coming off study will be contacted by telephone or at routine clinic visits approximately every 3 months until 36 months from date the last subject is randomized into the study.
Incidence of adverse events, significant laboratory value changes form baseline and anti-AMG 102 antibody formation. | Subjects coming off study will be contacted by telephone or at routine clinic visits approximately every 3 months until 36 months from date the last subject is randomized into the study.
Cmax and Cmin for AMG 102; Cmax and AUC for epirubicin and cisplatin with or without AMG 102 | Subjects coming off study will be contacted by telephone or at routine clinic visits approximately every 3 months until 36 months from date the last subject is randomized into the study.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Doshi S, Loh E, Oliner K, Gisleskog PO, Perez Ruixo JJ, Zhang Y, Zhu M.Exposure survival modeling.Journal-001088;
- [Background] Iveson T, Donehower RC, Davidenko I, Tjulandin S, Deptala A, Harrison M, Nirni S, Lakshmaiah K, Thomas A, Jiang Y, Zhu M, Tang R, Anderson A, Dubey S, Oliner KS, Loh E. Rilotumumab in combination with epirubicin, cisplatin, and capecitabine as first-line treatment for gastric or oesophagogastric junction adenocarcinoma: an open-label, dose de-escalation phase 1b study and a double-blind, randomised phase 2 study. Lancet Oncol. 2014 Aug;15(9):1007-18. doi: 10.1016/S1470-2045(14)70023-3. Epub 2014 Jun 22. PMID 24965569
- [Background] Oliner K.BM Ph2 Gastric.Journal-004521;
- [Background] TBD.Ph2 Gastric Exposure Response.Journal-004521;
- [Background] TBD.Ph2 Gastric PRO.Journal-004521;
- [Background] Zhu.20060317 ER data.Journal-000728;
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com